CLINICAL TRIAL: NCT04849728
Title: A Randomised, Double-blind, Placebo-controlled, Multicentre, Phase 3 Study Evaluating Efficacy and Safety of Lanifibranor Followed by an Active Treatment Extension in Adult Patients With Non-cirrhotic Non-alcoholic Steatohepatitis (NASH) and Fibrosis Stages F2 and F3
Brief Title: A Phase 3 Study Evaluating Efficacy and Safety of Lanifibranor Followed by an Active Treatment Extension in Adult Patients With (NASH) and Fibrosis Stages F2 and F3 ( NATiV3 )
Acronym: NATiV3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inventiva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 337HNAS20011
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Phase III; Nonalcoholic Steatohepatitis; NASH; Peroxisome proliferator-activated receptor (PPAR); Liver Diseases; Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fibrosis | interventions — lanifibranor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lanifibranor (IVA 337) (800 mg/day) (Experimental): 2 Lanifibranor tablets 400mg + 1 Placebo to match tablet with food --> once a day (quaque die, QD)
  Interventions: Drug: IVA337; Drug: Placebo
- Lanifibranor (IVA 337) (1200 mg/day) (Experimental): 3 Lanifibranor tablets 400mg with food --> once a day (quaque die, QD)
  Interventions: Drug: IVA337
- Matching placebo (Placebo Comparator): 3 Placebo to match tablets with food --> once a day (quaque die, QD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IVA337 — A total of 1000 patients will be randomised to receive lanifibranor (800 mg/day) or lanifibranor (1200 mg/day), or matching placebo, employing a 1:1:1 randomisation scheme, respectively, without interruption between Part A and Part B.
  Other Names: Lanifibranor
  Arms: Lanifibranor (IVA 337) (1200 mg/day); Lanifibranor (IVA 337) (800 mg/day)
Drug: Placebo — A total of 1000 patients will be randomised to receive lanifibranor (800 mg/day) or lanifibranor (1200 mg/day), or matching placebo, employing a 1:1:1 randomisation scheme, respectively, without interruption between Part A and Part B.
  Arms: Lanifibranor (IVA 337) (800 mg/day); Matching placebo

SUMMARY:
This Phase 3 study is conducted to evaluate lanifibranor in adults with NASH and liver fibrosis histological stage F2 or F3

DETAILED DESCRIPTION:
Primary objectives

This Phase 3 study is conducted to evaluate lanifibranor in adults with NASH and liver fibrosis stage F2 or F3 and consists of 2 sequential parts - an initial double-blind placebo-controlled (DBPC) period (Part A) followed by a double-blind active treatment extension (ATE) period (Part B), with the following primary objectives:

Part A To assess the safety and efficacy of lanifibranor compared to placebo on 'NASH resolution and improvement of fibrosis' assessed by liver histology.

Part B To assess the safety of lanifibranor beyond the DBPC period. Secondary objectives

Key secondary objectives of Part 1:

* To assess the effect of lanifibranor compared to placebo on NASH resolution and no worsening of fibrosis
* To assess the effect of lanifibranor compared to placebo on improvement of fibrosis with no worsening of NASH

Other secondary objectives of both Part 1 and Part 2:

* To assess the effect of lanifibranor on other key histological features of NASH (only for DBPC period)
* To assess the effect of lanifibranor on NASH resolution and improvement of fibrosis in diabetic patients (only for DBPC period)
* To assess the effect of lanifibranor on liver tests
* To assess the effect of lanifibranor on glycaemic parameters
* To assess the effect of lanifibranor on lipid parameters
* To assess the effect of lanifibranor on liver stiffness and steatosis assessed by elastography.
* To assess the effect of lanifibranor on health-related quality of life
* To assess the safety of lanifibranor
* To assess population PK modeling through plasma levels of lanifibranor using sparse sampling scheme (only for DBPC period)

ELIGIBILITY:
Prescreening Criteria:

* Diagnosed with NASH on prior liver biopsy
* Type 2 diabetes with high waist circumference or obesity or hepatic steatosis on ultrasound
* At least 3 of the components of metabolic syndrome

Inclusion Criteria:

1. Male or female, aged ≥18 years at the time of signing informed consent
2. Upon central biopsy reading process: diagnosis of NASH according to the Steatosis-Activity-Fibrosis (SAF):

   1. Steatosis score ≥1
   2. Activity score: A3 or A4
   3. Fibrosis score: F2 or F3
3. No qualitative change in dose for the drugs listed below:

   1. Antidiabetic treatment if glucagon-like peptide-1 receptor agonists (GLP1 receptor agonists) or sodium-glucose co-transporter-2 inhibitors (SGLT2 inhibitors): for at least 3 months
   2. Vitamin E (if at a dose ≥400 IU/day): for at least 6 months
   3. Statins: for at least 3 months
4. No qualitative change in dose for all other chronically administered drugs for at least 3 months prior to Screening
5. Weight stable for 6 months prior to Screening and between the qualifying liver biopsy and Baseline (no more than 5% change for both periods)
6. Negative serum pregnancy test at study Screening for females of childbearing potential confirmed by central laboratory. Females of childbearing potential must practice a consistent and proper use of highly effective method of contraception throughout the study and for 1 month after treatment discontinuation.

Exclusion Criteria:

Liver-related:

1. Documented causes of chronic liver disease other than NASH
2. Histologically documented liver cirrhosis (fibrosis stage F4)
3. History or current diagnosis of hepatocellular carcinoma (HCC)
4. History of or planned liver transplant
5. Positive human immunodeficiency virus (HIV) serology
6. ALT or AST >5 × ULN
7. AST<0.6 ULN if the liver biopsy has to be performed in the scope of the study
8. Abnormal synthetic liver function as defined by Screening central laboratory evaluation
9. Haemoglobin <110 g/L (11 g/dL) for females and <120 g/L (12 g/dL) for males
10. Patient currently receiving any approved treatment for NASH or obesity
11. Current or recent history (<5 years) of significant alcohol consumption
12. Treatment with drugs that may cause non-alcoholic fatty liver disease (NAFLD) administered for at least 2 weeks within 12 months prior to qualifying liver biopsy

    Glycaemia related:
13. HbA1c >9% at Screening
14. Diabetes mellitus other than type 2
15. Current treatment with insulin
16. Treatment with PPAR-gamma agonists (thiazolidinediones [TZDs]) 12 months before screening or historical biopsy.

    Obesity related:
17. Bariatric surgery: Restrictive procedures are allowed, if performed >6 months prior to the qualifying liver biopsy; malabsorptive procedures and procedures combining both restrictive and malabsorptive methods are not allowed within 5 years of the qualifying liver biopsy.

    Cardiovascular related:
18. History of heart failure with reduced left ventricular ejection fraction (LVEF)
19. Atrial fibrillation requiring anticoagulation
20. Unstable heart failure
21. Uncontrolled hypertension at Screening (values >160/100 mm Hg)

    General safety:
22. Women currently breastfeeding
23. Previous exposure to lanifibranor
24. Participation in any clinical trial investigational medicinal product/device within 3 months from Screening or 5 half-lives from Screening, whichever is longer
25. Concomitant treatment with PPAR-alpha agonists (fibrates)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Resolution of NASH and improvement of fibrosis | Part A: Date of randomisation until the date of biopsy at Week 72
  Part A: DBPC: Resolution of NASH and improvement of fibrosis at Week 72, defined by NASH CRN scores for ballooning of 0 and inflammation of 0 to 1, and fibrosis score ≥1 stage decrease compared to Baseline
Safety Analyses | 48 weeks after completion of DBPC period
  Part B: ATE:
  * Using the DBPC on-treatment period, comparing the 2 active arms versus placebo
  * Using the DBPC +ATE on treatment periods, assessing the 2 active arms. For adverse events, adjudicated liver events, and DILI and MACE events, in addition to the raw cumulative incidence proportions, the exposure-adjusted incidence rates will be provided based on the time patients are at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Arun J Sanyal, MD, Principal Investigator — VCU Health, Gastroenterology Hepatology and Nutrition, 1200 West Broad Street, Richmond VA23298, USA; Sven Francque, MD, Principal Investigator — Division of Gastroenterology and Hepatology, Antwerp University Hospital, Wilrijkstraat 10, B-2650 Edegem, Belgium
Locations (487):
- United States (223):
  - Pinnacle Research Group, Anniston, Alabama
  - Objective Health - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Digestive Health Specialist of the Southeast, Dothan, Alabama
  - North Alabama GI Research Center llc, Madison, Alabama
  - The Institute For Liver Health - Chandler, Chandler, Arizona
  - Arizona Liver Health - Peoria, Peoria, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Digestive Health - Sun City, Tucson, Arizona
  - Adobe Gastroenterology, Tucson, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Del Sol Research Management - Tucson East, Tucson, Arizona
  - ARcare Center for Clinical Research - Conway, Conway, Arkansas
  - ARcare Center for Clinical Research, Little Rock, Arkansas
  - Arkansas Diagnostic Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Office of Franco Felizarta, MD, Bakersfield, California
  - Fomatmedicalresearch, Camarillo, California
  - Precision Research Institute, Chula Vista, California
  - GW Research, Chula Vista, California
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - TriWest Research Associates, El Cajon, California
  - Cure Clinical Research, LLC, Fountain Valley, California
  - SC Clinical Research, Garden Grove, California
  - National Research Institute - Santa Ana, Huntington Park, California
  - The Clinical Trials Network - Gastro Care Institute, Lancaster, California
  - National Research Institute - Westlake, Los Angeles, California
  - National Research Institute - Panorama City, Panorama City, California
  - California Liver Reearch, Pasadena, California
  - Cadena Care Institute, Poway, California
  - Prospective Research Innovations Inc., Rancho Cucamonga, California
  - Stanford University Medical Center, Redwood City, California
  - Inland Empire Liver Foundation, Rialto, California
  - Research and Education, Inc., San Diego, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - Clinical Trial Management Services, Thousand Oaks, California
  - San Fernando Valley Health Institute, Van Nuys, California
  - South Denver Gastroenterology - Swedish Medical Center Office, Englewood, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - MedBio Trials, Adventura, Florida
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Synergy Healthcare, Bradenton, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Gastro Florida, Clearwater, Florida
  - Hi Tech and Global Research, LLC, Coral Gables, Florida
  - American Research Institute, INC, Cutler Bay, Florida
  - JY Research Institute Inc., Cutler Bay, Florida
  - Top Medical Research, Cutler Bay, Florida
  - Doral Medical Research, LLC, Hialeah, Florida
  - Palmetto Research, Hialeah, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Galenus Group, Lehigh Acres, Florida
  - Accel Research Sites, Maitland, Florida
  - Centor for Advanced Gastroenterology - Main Office - Maitland, Maitland, Florida
  - Florida Vascular Research, Miami, Florida
  - Life Medical Research Group, Miami, Florida
  - Optimus U Corporation, Miami, Florida
  - Schiff Center for Liver Diseases, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - USPA Advance Concept Medical Research Group, Miami, Florida
  - Future Care Solution, Miami, Florida
  - Genoma Research Group, Miami, Florida
  - Gastro Health - Galloway, Miami, Florida
  - Pro Live Medical Research, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Clinical Trials Services Corporation, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Sensible Healthcare Clinical Research, Ocoee, Florida
  - AdventHealth Transplant Institute, Orlando, Florida
  - Digestive and Liver Center of Florida - Orlando, Orlando, Florida
  - IMIC Research - International Medical Investigations Centers, Palmetto Bay, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - Pensacola GI Research Center, Pensacola, Florida
  - Eminat, LLC, Plantation, Florida
  - NAPA Research, Pompano Beach, Florida
  - Covenant Metabolic Specialists LLC - Sarasota, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - GI Alliance - Gastroenterology Associates of Florida - Wellington, Wellington, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Florida Medical Clinic - Zephyrhills, Zephyrhills, Florida
  - Athens Gastroenterology Association, Athens, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Research and Education Foundation of Atlanta Medical Center, Atlanta, Georgia
  - Oracle Clinical Research, College Park, Georgia
  - IACT Health, Columbus, Georgia
  - Southeast Clinical Research Center, Dalton, Georgia
  - Regional Infectious Diseases and Infusion Center, La Grange, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - ASHA Clinical Research - Munster, Hammond, Indiana
  - Heartland Medical Research, Clive, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Arizona Digestive Health - Sun City, Kansas City, Kansas
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Kansas Medical Clinic - Gastroenterology, Topeka, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Gastroenterology Associates - Baton Rouge, Baton Rouge, Louisiana
  - Tandem Clinical Research GI, Houma, Louisiana
  - Combined Gastro Research LLC, Lafayette, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Metropolitan Gastroenterology Associates - Metairie, Metairie, Louisiana
  - Tandem Clinical Research GI, LLC, Metairie, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Investigative Clinical Research - Annapolis, Annapolis, Maryland
  - Mercy Medical Center - Mcauley Plaza, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Digestive Disease Associates - Catonsville, Catonsville, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland - Columbia, Columbia, Maryland
  - Mid-Atlantic GI Research, Greenbelt, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Liver Center, Boston, Massachusetts
  - NECCR Prima Care Research, LLC, Fall River, Massachusetts
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - University of Michigan Health-West Hospital, Wyoming, Michigan
  - MNGI Digestive Health - Northeast Minneapolis Clinic, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Gastrointestinal Associates & Endoscopy Center - Flowood, Flowood, Mississippi
  - SKYCRNG - Quinn Healthcare, Ridgeland, Mississippi
  - Galen Research, Chesterfield, Missouri
  - Gastrointestinal (GI) Associates L.L.P., Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Sierra Clinical Research - Las Vegas, Las Vegas, Nevada
  - Southwest Gastroenterology Associates, Albuquerque, New Mexico
  - State University of New York - University at Buffalo, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Tandem Clinical Research - New York Clinic, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond University Medical Center, Staten Island, New York
  - Charlotte Gastroenterology and Hepatology - Randolph Road Office, Charlotte, North Carolina
  - ObjectiveGI - Northeast GI Research, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Gastroenterology of the Piedmont, PA - Salem Office, Winston-Salem, North Carolina
  - Consultants for Clinical Research - Montgomery Office, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Aventiv Research - Columbus, Columbus, Ohio
  - Digestive Specialists - Dayton, Dayton, Ohio
  - Ohio Gastroenterology Group, Inc. - Olentangy Office, Dublin, Ohio
  - Great Lakes Gastroenterology Research - Mentor, Mentor, Ohio
  - North Shore Gastroenterology, Westlake, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Options Health Research, Tulsa, Oklahoma
  - Veterans Affairs Pittsburgh Healthcare System - University Drive Campus, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Clinovacare Medical Clinical Research Center, West Columbia, South Carolina
  - Rapid City Medical Center, Rapid City, South Dakota
  - Gastro One - Germantown Office - Wolf Park Drive, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Accelemed Research Institute, Austin, Texas
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - South Texas Research Institute - Brownsville, Brownsville, Texas
  - PanAmerican Clinical Research - US Headquarters, Brownsville, Texas
  - Velocity Clinical Research - Austin, Cedar Park, Texas
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - GI Alliance - Texas Digestive Disease Consultants - Fort Worth - Downtown, Dallas, Texas
  - Soma Clinical Trials, Denison, Texas
  - South Texas Research Institute - Edinburg, Edinburg, Texas
  - Gastro Clinic, El Paso, Texas
  - Care United Medical Center - Forney, Forney, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Allure Health, Llc, Friendswood, Texas
  - Digestive Health Associates of Texas - Rockwall, Garland, Texas
  - Summitt - Pinnacle Clinical Research - Georgetown, Georgetown, Texas
  - Advanced Medical Trials, Georgetown, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Liver Associates of Texas, Houston, Texas
  - Liver Specialists of Texas, Houston, Texas
  - Gastroenterology Consultants - Ellington, Houston, Texas
  - Alpha Research Institute, LLC, Houston, Texas
  - Houston Research Institute (HRI), Houston, Texas
  - Headlands - Centex Studies - Westfield, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - GI Alliance - Lubbock Digestive Disease Associates - Lubbock, Lubbock, Texas
  - GI Alliance - Mansfield, Mansfield, Texas
  - Koncord Research - McAllen LLC, McAllen, Texas
  - Koncord Research-McAllen LLC, McAllen, Texas
  - Quality Research - San Antonio, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Texas Liver Institute/American Research Corporation, San Antonio, Texas
  - University of California San Diego, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Impact Research Institute, Waco, Texas
  - Digestive Health Research of Central Texas, Waco, Texas
  - GI Alliance - Bay Area Gastroenterology - Webster, Webster, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Digestive Health Research of North Texas, Wichita Falls, Texas
  - Lone Peak Family Health, Draper, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Inova Medical Group - Fairfax Hospital, Falls Church, Virginia
  - Emeritas Research Group, Leesburg, Virginia
  - Topography Health, Inc., Manassas, Virginia
  - Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - Digestive & Liver Disease Specialists, Norfolk, Virginia
  - GI Select Health Research, LLC, Richmond, Virginia
  - Hunter Holmes Mcguire Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano La Plata, La Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital De Alta Complejidad en Red El Cruce, Buenos Aires, Buenos Aries
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - Hospital Británico de Buenos Aires, Buenos Aires
- Australia (12):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Campbelltown Hospital, Liverpool, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Eastern Health - Australia, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Medizinische Universität Innsbruck, Innsbruck, Tyrol, Austria
- Belgium (11):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Hôpital Erasme, Brussels, Brussels Capital
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk, Limburg
  - Algemeen Ziekenhuis Maria Middelares, Ghent, Oost-Vlaaderen
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Vitaz, Sint-Niklaas, Oost-Vlaanderen
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
  - Algemeen Ziekenhuis Delta - Campus Rumbeke, Roeselare, West-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire de Liège Site Sart Tilman, Liège
- Brazil (6):
  - Hospital das Clinicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Ernesto Dornelles, Porto Alegre, Rio de Janeiro
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, Cerqueira César, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
- Bulgaria (7):
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N.I. Pirogov, Sofia, Sofia-Grad
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - Diagnostic Consultative Center Aleksandrovska, Sofia
  - Diagnostic Consulting Center 20 - Sofia Еооd, Sofia
  - Nov Rehabilitatsionen Tsentar EOOD, Stara Zagora
  - Medical Center Medica Plus, Veliko Tarnovo
- Canada (7):
  - Heritage Medical Research Centre, Calgary, Alberta
  - William Osler Health System - Brampton Civic Hospital, Brampton, Ontario
  - St. Joseph's Healthcare Hamilton - Charlton Campus, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Centre de Médecine Métabolique de Lanaudière, Terrebonne, Quebec
- Chile (3):
  - Hospital San Juan de Dios de La Serena, La Serena, Coquimbo Region
  - Centro De Investigaciones Clínicas Viña Del Mar, Viña del Mar, Región de Valparaíso
  - Pontificia Universidad Católica de Chile - Escuela de Medicina, Santiago
- China (61):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing university three gorges hospital, Chongqing, Chongging
  - First Affiliated Hospital of the Army Military Medical University (Southwest Hospital), Chongqing, Chongging
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Beijing You'an Hospital,Capital Medical University, Beijing, Fengtai
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Eighth Affiliated Hospital,GuangZhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Henan Provincal People's Hospital, Zhengzhou, Henan
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhengzhou First People's Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The Sixth People' s Hospital Of ShenYang, Shenyang, Liaoning
  - Xi'an International Medical Center, Xi'an, Shaanxi
  - Qingdao Central Hospital, Qingdao, Shandong
  - Xu, Jun The First Hospital of Shanxi Medical University Taiyun Shanxi, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan Shi
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital , Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - RuiAn People's Hospital - Ruixiang Branch, Ruian, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital - Central South University, Changsha
  - West china hospital Sichuan University, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Second Affiliated Hospital of Dalian Medical University, Dalian
  - Mengchao Hepatobiliary Hospital of FuJian Medical University, Fuzhou
  - Guangdong Provincial people's hospital, Guangzhou
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine - Qingchun Campus, Hangzhou
  - General Hospital of Tianjin Medical University, Heping
  - Ningbo No.2 Hospital (Hwa Mei Hospital), Ningbo
  - Qingdao Municipal Hospital, Qingdao
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - Tianjin Third Central Hospital, Tianjin
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhengzhou People's Hospital, Zhengzhou
- Czechia (2):
  - Research Site s.r.o., Pilsen
  - Synexus Czech - DRS Prague, Prague
- France (25):
  - Hôpital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - Hôpital Hautepierre, Strasbourg, Bas-Rhin
  - Hôpital Saint-Joseph, Marseille, Bouches-du-Rhône
  - CHU Dijon Bourgogne - Hôpital François Mitterrand, Dijon, Cantal
  - CHRU de Besançon - Hôpital Jean-Minjoz, Besançon, Franche-Comté
  - CHU de Lille - Hôpital Claude Huriez, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Rennes, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble, Isère
  - CHU de Limoges, Limoges, Limousin
  - Centre Hospitalier Universitaire De Nantes - Hôpital Nord Laennec, Nantes, Loire Atlantique
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Lorraine
  - Centre Hosptitalier Universitaire d'Angers, Angers, Maine-et-Loire
  - Centre Hospitalier Universitaire De Nantes - Hôpital Nord Laennec, Nantes, Nantes Cedex 1
  - Hôpital Haut-Lévêque, Pessac, Nouvelle-Aquitaine
  - CHU Saint-Eloi, Montpellier, Occitanie
  - Hôpital Rangueil, Toulouse, Occitanie
  - Clinique Pasteur, Toulouse, Occitanie
  - Hôpital l'Archet, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Puy-de-Dôme
  - Hôpital Cochin, Paris
  - Hôpitaux Universitaires Paris Nord Val-de-Seine - Hôpital Beaujon, Clichy, Île-de-France Region
  - Hôpitaux Universitaires Henri Mondor, Créteil, Île-de-France Region
  - Hôpital Universitaire Pitié Salpêtrière, Paris, Île-de-France Region
  - Hôpital Saint-Antoine, Paris, Île-de-France Region
  - Hôpitaux Universitaires Paris-Sud - Hôpital Paul Brousse, Villejuif, Île-de-France Region
- Germany (14):
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe, Baden-Wurttemberg
  - St. Josefs-Hospital Wiesbaden, Wiesbaden, Hesse
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Klinikum Chemnitz, Chemnitz, Saxony
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Eugastro, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
  - EPIMED, Berlin
  - Gastroenterologie am Bayerischen Platz, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Düsseldorf, Northeim
- Hungary (6):
  - SYNEXUS Magyarország Egészségügyi Szolgáltató KFT, Budapest, Central Hungary
  - Synexus Magyarország Egészségügyi Szolgáltató Kft. - Debrecen, Debrecen, Hajdú-Bihar
  - Debreceni Egyetem Klinikai Központ Kenézy Gyula Campus, Debrecen, Hajdú-Bihar
  - MIND Klinika, Budapest
  - High Tech Medical Kft., Budapest
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest
- Israel (8):
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Gush Dan
  - Carmel Medical Center, Haifa, Haifa District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem, Jerusalem
  - Western Galilee Hospital-Nahariya, Nahariya, Northern District
  - Soroka Medical Center, Beersheba, Southern District
  - The Chaim Sheba Medical Center, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus, Haifa
- Italy (10):
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milan
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Università degli Studi di Napoli Federico II, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - UOSD Interdipartimentale Degenza Medica a ciclo breve, Roma
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino
- Mexico (18):
  - Centro de Investigacion Medico Biologica y Terapia Avanzada, Guadalajara, Jalisco
  - Centro de Investigación y Gastroenterología, Cuauhtémoc, Mexico City
  - PanAmerican Clinical Research Mexico - Cuernavaca, Cuernavaca, Morelos
  - Investigaciones Medicas Cisneros, Monterrey, Nuevo León
  - Hospital Universitario Doctor José Eleuterio Gonzalez, Monterrey, Nuevo León
  - Medical Care and Research S.A. de C.V., Mérida, Yucatán
  - Consultorio de la Dra. Maria Sarai Gonzalez Huezo, Metepec
  - Instituto de Seguridad Social del Estado de Mexico y Municipios, Metepec
  - Oaxaca Site Management Organization S.C., Metepec
  - Centro de Investigacion y Gastroenterologia, S.C., Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ), Mexico City
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" (Servicio de Gastroenterologia), Monterrey
  - Hospital Universitario "Dr. José Eleuterio González" (Servicio de Endocrinología), Monterrey
  - Hospital Universitario Dr. José Eleuterio González, Monterrey
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - PanAmerican Clinical Research S.A. de C.V., Querétaro
  - Hospital Regional de Alta Especialidad de Zumpango, Zumpango
- Netherlands (7):
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Ziekenhuis Bernhoven, Uden, North Brabent
  - Amsterdam Universitair Medische Centra - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (11):
  - Synexus - Poznań, Poznan, Greater Poland Voivodeship
  - Synexus - Wrocław, Wroclaw, Lower Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Badan Klinicznych, Wroclaw, Lower Silesian Voivodeship
  - Synexus - Warszawa, Warsaw, Masovian Voivodeship
  - Synexus - Gdynia, Gdynia, Pomeranian Voivodeship
  - Synexus - Częstochowa, Częstochowa, Silesian Voivodeship
  - Synexus - Katowice, Katowice, Silesian Voivodeship
  - Centrum Medyczne Pratia - Katowice, Katowice, Silesian Voivodeship
  - ID Clinic, Mysłowice, Silesian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus - Łódź, Lodz, Łódź Voivodeship
- Portugal (7):
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães, Braga District
  - Hospital de Braga, Braga
  - Centro Hospitalar Universitário Lisboa Norte - Hospital De Santa Maria, Lisbon
  - Centro Hospitalar Universitário De São João, Porto
  - Hospital Pedro Hispano, Senhora da Hora
  - Unidade Local Saúde Alto Minho - Hospital de Santa Luzia, Viana do Castelo
  - Centro Hospitalar de Trás-Os-Montes e Alto-Douro - Hospital de S. Pedro, Vila Real
- Fundación de Investigación de Diego Clinical Research, San Juan, Puerto Rico
- South Africa (4):
  - Sefako Makgatho Health Sciences University, Pretoria, Gauteng
  - Synexus - Mediclinic Southern Africa - Constantiaberg, Cape Town, Western Cape
  - Synexus - Helderberg Clinical Research Centre - Somerset West, Somerset West, Western Cape
  - Synexus Clinical Research SA- Watermeyer, Pretoria
- Spain (23):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Complejo Asistencial Universitario de Leon, León
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clínica Universidad de Navarra, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complejo Hospitalario De Pontevedra, Pontevedra
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Consorci Hospital General Universitari de València, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Ukraine (3):
  - Medical Center Edelweiss Medics, LLC, Kyiv
  - Medical Center Medbud-Clinic, LLC, Kyiv
  - Medical Center Center of Family Medicine Plus, LLC, Kyiv
- United Kingdom (11):
  - Barts Health NHS Trust, London, England
  - Panthera Biopartners - North London, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Panthera Biopartners - Manchester, Manchester, England
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Panthera Biopartners - Preston, Preston, England
  - Sheffield Teaching Hospitals NHS FT, Sheffield, England
  - Royal Surrey County Hospital NHS Foundation Trust, Surrey Quays, England
  - Panthera Biopartners - Glasgow, Glasgow, North Lanarkshire
  - Royal Free London NHS Foundation Trust, London